CLINICAL TRIAL: NCT01274091
Title: Gene-diet Interactions
Brief Title: Gene - Diet Interactions
Acronym: Genediet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 28//2010
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Insulin Sensitivity
Keywords: Gene-diet interaction; PPARgamma gene; Pro12Ala; Fatty acids; Dietary modification; Insulin sensitivity; Glucose metabolism
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- P/S-ratio 1.0 (Experimental): Diets will contain 30% of energy as fat, 18% as protein and 52% as carbohydrates:
  polyunsaturated fatty acid diet (PUFA) will have P/S ratio 1.0.
  Interventions: Other: PUFA-diet
- P/S-ration 0.3 (Experimental): Diets will contain 30% of energy as fat, 18% as protein and 52% as carbohydrates:. Saturated fatty acid diet (SAFA) will polyunsaturated/saturated (P/S) ratio of 0.3.
  Interventions: Other: SAFA-diet

INTERVENTIONS:
Other: PUFA-diet — Diets will contain 30% of energy as fat, 18% as protein and 52% as carbohydrates: polyunsaturated fatty acid diet (PUFA) will have P/S ratio 1.0.
  Arms: P/S-ratio 1.0
Other: SAFA-diet — Diets will contain 30% of energy as fat, 18% as protein and 52% as carbohydrates: Saturated fatty acid diet (SAFA) will polyunsaturated/saturated (P/S) ratio of 0.3.
  Arms: P/S-ration 0.3

SUMMARY:
Interactions between genes and environment, i.e. our inherited responses to environmental changes, may be crucial in the development of the common diseases. The investigators were the first to identify PPARG gene as risk gene for type 2 diabetes. The role of the Pro12Ala polymorphism in diabetes risk has also been verified in meta-analysis. However, this effect on seems to depend on intervention and age. In this study the effects of diets high with saturated fatty acids (SAFA) and polyunsaturated fatty acids (PUFA) are compared in subjects carrying either Pro12Pro or Ala12Ala genotype of the PPARG gene.

Aim of the study:

To test if subjects with Pro12Pro and Ala12Ala genotypes respond differentially to a diet supplemented with high saturated (SAFA) or polyunsaturated fat (PUFA).

Hypotheses:

1. Specific: Subjects with the Ala12Ala genotype will be more sensitive to dietary modification, and therefore respond more favorably to PUFA diet
2. More general: Dietary instructions individually tailored according to the genotype would allow better treatment of obesity and diabetes

DETAILED DESCRIPTION:
Obesity and type 2 diabetes are increasing in all western countries, including Finland. Recent genome wide analyses have found > 30 genes that contribute to either condition.. However, none of these genes explain >5% of the disease risk and altogether they explain < 10% of the total disease risk in cross-sectional studies. Therefore, diet and physical activity are still the major determinants of the risk, as demonstrated by our earlier intervention studies in order to find out the effect of different dietary modifications on glucose and lipid metabolism. More importantly, interactions between genes and environment, i.e. our inherited responses to environmental changes, may be crucial in the development of the common diseases. Unfortunately, gene-environment interaction can only be effectively investigated in intervention studies that are more expensive than cross-sectional population screenings. This leads to a lower sample size and reduced power to detect effects of minor alleles. Despite these limitations the investigators have been able to demonstrate gene-intervention interactions for several genes, including PPARG, in the Finnish Diabetes Prevention study. There is an urgent need for studies investigating effects of tailored diets in individuals selected based on their genotype. This will be the next essential step leading to improved dietary treatments guided by genetic information.

The investigators were the first to identify PPARG gene as risk gene for type 2 diabetes. The role of the Pro12Ala polymorphism in diabetes risk has also been verified in meta-analysis. However, this effect on seems to depend on intervention and age. Based on these findings the investigators created in collaboration with Johan Auwerx an Pro12Ala animal model that demonstrated a differential effect of dietary fat composition depending on the genotype. However, an important conclusive proof that subjects selected based on their Pro12Ala genotype would respond differently to specifically tailored diet modification is still needed.

In this study the effects of diets high with saturated fatty acids (SAFA) and polyunsaturated fatty acids (PUFA) are compared in subjects carrying either Pro12Pro or Ala12Ala genotype of the PPARG gene. As a primary endpoint the investigators expect insulin sensitivity to alter differently depending on the genotype. Additionally, a detailed characterization of energy, glucose and lipid metabolism will be performed. Because PPARG gene plays a central role in adipogenesis one of the aims of this study is to find new pathways, genes and gene clusters that are regulated by PPARG in humans.

ELIGIBILITY:
Inclusion Criteria:

* BMI >20kg/m2 <29kg/m2
* Pro12Pro and Ala12Ala genotypes of PPARG Pro12Ala polymorphism
* participation to METSIM-study (METabolic Syndrome in Men, currently >10000 men included from the population living in Kuopio, principal investigator Markku Laakso)
* normoglycemia

Exclusion Criteria:

* type 2 diabetes
* other chronic diseases

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | week 0
  insulin sensitivity measured by oral glucose tolerance test at the beginning of the first, randomised diet
insulin sensitivity | week 8
  insulin sensitivty measured by oral glucose tolerance test after the first diet
insulin sensitivity | week 10
  Insulin sensitivity measured by oral glucose tolerance test in the beginning of the second, randomised diet
insulin sensitivity | week 18
  insulin sensitivity measured by oral glucose tolerance test after the second diet

SECONDARY OUTCOMES:
peripheral blood mononuclear cell gene expression | week 8
peripheral blood mononuclear cell gene expression | week 18
serum lipids | week 8
  serum lipids, including serum lipidomics and fatty acid composition
serum lipids | week 18
  serum lipids, including serum lipidomics and fatty acid composition
inflammation | week 8
  inflammation measured as serum cytokines and adipose tissue inflammation
inflammation | week 18
  inflammation measured as serum cytokines and adipose tissue inflammation
energy expenditure | week 8
  energy expenditure and the rates of substrate oxidation
energy expenditure | week 18
  energy expenditure and the rates of substrate oxidation
insulin secretion | week 8
insulin secretion | week 18
adipose tissue gene expression | week 8
adipose tissue gene expression | week 18

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Pihlajamäki, Professor, Principal Investigator — University of Eastern Finland, Kuopio University Hospital; Ursula S Schwab, Clinical Lect, adjunct prof, Study Director — University of Eastern Finland; Matti Uusitupa, Professor, Study Chair — Professor
Locations (1):
- University of Eastern Finland, Kuopio, Finland